CLINICAL TRIAL: NCT03541642
Title: Development and Pilot Testing of a PrEP Communication Intervention and Integration Into Existing HIV Testing Services for Female IV Drug Using Clients of a Needle Exchange
Brief Title: PrEP Communication Intervention for Female Clients of a Needle Exchange
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25028
Record Dates: First submitted 2018-02-28; First posted 2018-05-30 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Women participants will be randomized to condition upon consent based on a random numbers table. Intervention arm will get "enhanced" intervention with customized messages and counseling/text messaging; control arm will get "basic" intervention with medical counseling and text message reminders.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Intervention (Experimental): Women who are eligible and randomized to the Enhanced Intervention will receive targeted PrEP counseling; targeted written/visual materials, follow up supportive text messages, and distribution of PrEP at the syringe exchange
  Interventions: Behavioral: Enhanced Intervention
- Basic Intervention (Active Comparator): Women who are eligible and randomized to the Basic Intervention will receive "usual care" with general messaging from medical personnel, reminder text messages, and distribution of PrEP at the syringe exchange
  Interventions: Behavioral: Basic Intervention

INTERVENTIONS:
Behavioral: Enhanced Intervention — Targeted PrEP counseling; targeted written/visual materials; follow up supportive text messages; distribution of PrEP at the syringe exchange
  Arms: Enhanced Intervention
Behavioral: Basic Intervention — General messaging from medical personnel; reminder text messages; distribution of PrEP at the syringe exchange
  Arms: Basic Intervention

SUMMARY:
This study will identify perceptions of PrEP in women who inject drugs (WWIDs) and develop and pilot test a targeted intervention that will be embedded in a large, urban syringe exchange program through an extensive formative evaluation process. Using perceptual mapping, an innovative marketing evaluation technique, WWIDs' PrEP perceptions will be incorporated into messaging in targeted counseling, materials, and text messaging to encourage PrEP adherence. This will then be tested in a pilot Randomized Controlled Trial (RCT) by comparing it to a general PrEP intervention to assess for uptake and adherence to PrEP, as well as improved self-efficacy and lower decisional conflict.

DETAILED DESCRIPTION:
Women who inject drugs (WWIDs) are at significantly higher risk of contracting HIV due to both needle sharing and sexual behaviors, yet utilize HIV prevention resources less. Analysis of studies testing pre-exposure prophylaxis (PrEP) has not tested effectiveness in WWIDs and little research exists on their specific barriers to uptake and adherence. The result is a significant group who is highly vulnerable to HIV infection and its negative health consequences, yet is less likely to benefit from PrEP. To address this gap this study will use a rigorous formative evaluation strategy utilizing a unique and innovative marketing evaluation technique. Using perceptual mapping and vector modeling analysis, the investigators will develop 3-D maps to identify specific message strategies to embed into an intervention using targeted PrEP counseling, written materials, and text based messaging and pilot tested for promise of efficacy compared to a general PrEP intervention. The intervention will address psycho-social barriers to PrEP through perceptual mapping but also societal and structural barriers by embedding it in a trusted syringe exchange and distributing medication through its medical clinic. Specific aims of the research are: 1. Assess WWIDs' perceptions of PrEP and potential barriers to use. To accomplish this the investigators will conduct focus groups (n=30) and interviews with syringe exchange staff (n=10) and develop a perceptual mapping survey. 2. Develop a targeted communication intervention based on vector modeling findings, including print materials, PrEP counseling, and text messages, and assess feasibility and acceptability. To accomplish this the investigators will conduct perceptual mapping surveys with HIV- WWIDs (n=100), do vector modeling analysis and create sample messages, concept test messages with WWIDs and staff (n=20), create intervention materials and conduct usability testing (n=20). 3. Pilot test the intervention by integrating into a syringe exchange to assess promise of efficacy. To accomplish this the investigators will conduct a randomized pilot (n=50) and test an "enhanced" intervention using targeted messages with a "basic" intervention that provides general PrEP counseling. To assess promise of efficacy the investigators will compare PrEP adherence (blood test; self report) and differences in PrEP attitudes, self-efficacy, and decisional conflict.

ELIGIBILITY:
Inclusion Criteria:

* self-identifying women -HIV-
* 18 or older
* self-report either sharing needles or having unprotected sex in last month
* speak and read English
* Is not currently PrEP
* have cell phone that receives text messages
* have Medicaid/Medicare or other insurance that covers PrEP

Exclusion Criteria:

* self-identifying other than female
* HIV+
* under 18 years old
* Doesn't speak/read English
* No HIV risk in last three months
* Are on PrEP
* Do not have a cell phone that accepts text messages
* Do not have insurance that covers PrEP
* mental illness that interferes with cognitive understanding or ability to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Any self-reported women who injects drugs or has other HIV risk related to drug use
Enrollment: 35 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah B Bass, PhD, MPH, Principal Investigator — Temple University
Locations (1):
- Prevention Point Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All research products from the study will be made available to other qualified individuals within the scientific community, government agencies and other interested parties after publication of results. Requests for raw data from other scientists will be considered with provision of the following information: A brief description of the specific aims and/or hypotheses, data requirements, and proposed analyses, how the data will be used, timeframe for use, and Institutional Review Board (IRB) approvals. All materials developed during the study, as well as any research instruments, will also be made available upon request. In addition, qualified individuals who are interested in the PrEP messaging and the methods from which they are created, as well as the analysis methods generated by this research, will have access after publication. It is our full intention to share all findings generated by this study, and subsequent lessons learned, with others in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Three months after end of intervention data collection.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited for the pilot clinical trial from September 2020 to September 2021. Participants were recruited for the formative work that was done prior to developing the intervention on June 1, 2018. All were self-identified females who were clients of Prevention Point Philadelphia, a social services agency and syringe services exchange.
Pre-assignment Details: A total of 35 participants were randomized to intervention or control arms. IRB required us to consent women prior to eligibility due to HIPAA. In total, forty nine women were recruited and 48 consented for the study prior to eligibility. Of these, 12 were found to be not eligible based on criteria (i.e. previously used PrEP, no reported HIV risk behavior, no phone). Of the 36 remaining, one was lost before randomization could occur, resulting in a final group of 35 participants.
Period: Overall Study
Arm/Group | Enhanced Intervention | Basic Intervention
Started | 19 | 16
1-month | 3 | 4
3-month | 1 | 3
3-month Follow-up | 1 | 1
Completed | 1 | 1
Not Completed | 18 | 15
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 16 | 12
Not completed — Found out previously on PrEP after randomization before eligibility was expanded | 1 | 1

BASELINE CHARACTERISTICS:
Population: The number of participants in the Baseline Analysis Population only includes participants who completed the baseline survey in its entirety. 35 participants were randomized to a condition. However, 2 participants were later deemed ineligible as they had previously taken PrEP. 2 additional participants did not complete the baseline assessment in its entirety. In total, 31 participants were randomized, eligible, and completed baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Intervention | Basic Intervention | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.24 (10.35) | 39.86 (8.54) | 40.06 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 12 | 8 | 20
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 31
Coping Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Assess coping self-efficacy using the Coping Self-Efficacy Scale (13 item scale; 0-10 scale). Zero=cannot do at all,5=moderately certain can do and 10=certain can do. An overall CSE score (from 0 to 130) is created by summing the item ratings, with higher scores indicating higher coping self-efficacy. Population: Analysis population only includes cases that completed baseline. Note that one item of the CSE scale was inadvertently excluded from the baseline measure. Random imputation was used to populate a value from 0-10 for this missing item value prior to scoring the CSE.
  units on a scale
    number analyzed (Participants) | 13 | 12 | 25
    (all) | 83.23 (15.85) | 87.83 (18.90) | 85.44 (17.17)
Decisional Conflict [Mean (Standard Deviation); unit: units on a scale] — Assess decisional conflict with the Ottawa Decisional Conflict Scale. 13 items. 5 responses: Strongly Disagree (1), Disagree (2), Neither Agree or Disagree (3), Agree (4), Strongly Agree (5). The scores on the 13 items were summed and then divided by the number of items (13) to produce an overall mean, ranging from 1 to 5. The lower the score, the lower the decisional conflict. A mean of 4 is considered higher decisional conflict.
  units on a scale | 4.35 (0.58) | 4.28 (0.48) | 4.32 (0.53)
PrEP Benefits [Mean (Standard Deviation); unit: units on a scale] — 10 items assessed perceived benefits of PrEP. Items are asked on a 0-10 Likert, with 0 = strongly disagree, 5 = unsure, 10 = strongly agree. Thus, higher score indicates greater agreement with that item.
  units on a scale
    PrEP can keep me from getting HIV | 9.06 (1.78) | 9.07 (1.21) | 9.06 (1.53)
    Using PrEP would make me feel more in charge of my life | 7.71 (3.35) | 8.36 (1.50) | 8.00 (2.66)
    I would be able to enjoy sex more if I was taking PrEP | 6.88 (3.33) | 6.43 (3.94) | 6.68 (3.33)
    PrEP is easy to take | 9.41 (1.33) | 9.79 (0.80) | 9.58 (1.12)
    PrEP would not interfere with me injecting or taking drugs | 9.00 (1.97) | 8.64 (2.10) | 8.84 (2.00)
    I would not have to rely on my partner to use condoms if I was taking PrEP | 2.12 (2.85) | 3.36 (3.78) | 2.68 (3.30)
    I would only have to take one pill a day if I was on PrEP | 9.18 (1.85) | 9.14 (1.56) | 9.16 (1.70)
    PrEP would let me worry less about HIV | 9.29 (1.36) | 8.07 (3.29) | 8.74 (2.46)
    I would not have to feel guilty about. having fun if I took PrEP | 5.41 (3.79) | 6.07 (3.95) | 5.71 (3.81)
    PrEP is affordable | 8.35 (2.74) | 8.36 (1.95) | 8.35 (2.37)
PrEP Barriers [Mean (Standard Deviation); unit: units on a scale] — 12 items assessed perceived barriers to taking PrEP. Items are asked on a 0-10 Likert, with 0 = strongly disagree, 5 = unsure, 10 = strongly agree. Thus, higher score indicates greater agreement with that item.
  units on a scale
    It would be hard for me to take a pill every day | 1.41 (2.62) | 1.93 (3.20) | 1.65 (2.86)
    Taking PrEP would dull my high | 0.59 (1.33) | 0.64 (1.50) | 0.61 (1.38)
    Taking PrEP would cause too many side effects | 1.41 (2.15) | 2.36 (2.41) | 1.84 (2.28)
    I feel healthy so I don't need to take PrEP | 1.12 (2.42) | 2.00 (3.35) | 1.52 (2.86)
    I already protect myself from HIV in other ways (i.e., condoms, not sharing needles) | 3.65 (4.00) | 4.29 (3.34) | 3.94 (3.67)
    Even if I take PrEP, I might get HIV anyway | 4.82 (4.07) | 5.50 (3.53) | 5.13 (3.78)
    PrEP only protects against HIV, not other sexually transmitted infections | 8.88 (2.45) | 8.71 (2.05) | 8.81 (2.24)
    My partner might hurt me if they knew I was on PrEP | 0.41 (1.28) | 0.86 (1.83) | 0.61 (1.54)
    I have a lot more worries in my life than getting HIV | 3.41 (3.97) | 3.86 (3.53) | 3.61 (3.72)
    If I started PrEP it would be hard to get to the doctor every three months | 0.82 (1.38) | 0.86 (1.70) | 0.84 (1.51)
    I don't have a safe place to keep PrEP | 1.71 (2.73) | 1.36 (2.87) | 1.55 (2.15)
    I would be afraid if I had PrEP it would get stolen | 1.59 (2.15) | 1.71 (2.84) | 1.65 (2.44)
PrEP Beliefs [Mean (Standard Deviation); unit: units on a scale] — 9 items assessed perceived beliefs about PrEP. Items are asked on a 0-10 Likert, with 0 = strongly disagree, 5 = unsure, 10 = strongly agree. Thus, higher score indicates greater agreement with that item. Population: One participant in the enhanced group did not provide a response to item "PrEP sounds too good to be true". Thus, the analysis population was reduced from 17 to 16.
  units on a scale
    Sex workers need PrEP more than other people | 5.29 (4.52) | 3.79 (3.45) | 4.61 (4.08)
    People who inject drugs need PrEP more than other people | 6.00 (4.11) | 4.79 (4.00) | 5.45 (4.04)
    Gay men need PrEP more than other people | 3.88 (3.48) | 3.64 (3.99) | 3.77 (3.66)
    Trans people need PrEP more than other people | 3.65 (3.55) | 3.29 (3.58) | 3.48 (3.51)
    People from certain races/ethnicities need PrEP more than other people | 1.65 (2.64) | 1.43 (2.17) | 1.55 (2.41)
    PrEP sounds too good to be true: number analyzed (Participants) | 16 | 14 | 30
    PrEP sounds too good to be true | 2.19 (3.43) | 2.14 (2.71) | 2.17 (3.06)
    PrEP makes people think they are invincible (can't get HIV or other sexually transmitted infections) | 2.12 (2.85) | 3.00 (3.66) | 2.52 (3.21)
    PrEP is safe and effective for women to use | 9.24 (1.35) | 8.43 (2.74) | 8.87 (2.09)
    I am more likely to take PrEP if I am being paid to take it | 2.71 (3.65) | 3.07 (3.69) | 2.87 (3.61)

OUTCOME MEASURES:

1. Primary Outcome: Change in PrEP Uptake and Adherence
Description: Self-report PrEP adherence and bio-verified PrEP adherence to PrEP with urine assay (Synergy medical labs - Descovy Panel TFV:Creatinine Ratio-Descovy). Urine assay results will be categorized as a binary variable (yes/no) based upon value observed by all patients, with data at 1 month, 3 months and 3 months post intervention.
Time Frame: one month, three months, three months post intervention
Population: The enhanced intervention group analysis population at 1 month (n=3) differs from the overall enhanced intervention group n (17), and basic intervention group analysis population at 1 month (n=4) differs from the overall basic intervention group n (14) due to implementation barriers that prevented women from getting onto PrEP (e.g., lack of venous access, not returning for doctor appointment), and remaining adherent (failure to pick up meds, failure to show for appointments).
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Intervention | Basic Intervention
Number analyzed (Participants) | 3 | 4
Participants
  1 month: Still taking PrEP, bio-verified | 0 | 1
  1 month: Still taking PrEP, not bio-verified | 2 | 3
  1 month: Not taking PrEP | 1 | 0
  3 month: number analyzed (Participants) | 1 | 3
  3 month: Still taking PrEP, bio-verified | 0 | 1
  3 month: Still taking PrEP, not bio-verified | 0 | 2
  3 month: Not taking PrEP | 1 | 0
  3 month follow up: number analyzed (Participants) | 1 | 1
  3 month follow up: Still taking PrEP, bio-verified | 0 | 0
  3 month follow up: Still taking PrEP, not bio-verified | 0 | 0
  3 month follow up: Not taking PrEP | 1 | 1

2. Primary Outcome: PrEP Adherence Within Past Week
Description: Self report PrEP adherence measure of PrEP use within the past week. Item asks "Of the seven doses of PrEP you were supposed to take during the last week, how many doses would you say you missed? Responses range from 0 to 7.
Time Frame: one month, three months, three months post intervention
Population: Enhanced group at 1month (n=3) differs from the overall enhanced group n (17) & basic group at 1 month (n=4) differs from overall basic group n (14) due to implementation barriers that prevented PrEP uptake (e.g., lack of venous access, not returning for doctor appointment), and remaining PrEP adherent (failure to pick up meds, failure to show for appointments). Drop off at 3 month is due to lost to follow up & dropout. No participant at 3 month follow up reported PrEP use.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Intervention | Basic Intervention
Number analyzed (Participants) | 3 | 4
Participants
  1 month: 7 days | 1 | 0
  1 month: 6 days | 0 | 0
  1 month: 5 days | 0 | 0
  1 month: 4 days | 0 | 0
  1 month: 3 days | 1 | 0
  1 month: 2 days | 1 | 0
  1 month: 1 day | 0 | 0
  1 month: 0 days | 0 | 4
  1 month: Unknown or not reported | 0 | 0
  3 month: number analyzed (Participants) | 1 | 3
  3 month: 7 days | 0 | 0
  3 month: 6 days | 0 | 0
  3 month: 5 days | 0 | 0
  3 month: 4 days | 0 | 0
  3 month: 3 days | 0 | 0
  3 month: 2 days | 0 | 0
  3 month: 1 day | 0 | 1
  3 month: 0 days | 0 | 2
  3 month: Unknown or not reported | 1 | 0
  3 month follow up: number analyzed (Participants) | 1 | 1
  3 month follow up: 7 days | 0 | 0
  3 month follow up: 6 days | 0 | 0
  3 month follow up: 5 days | 0 | 0
  3 month follow up: 4 days | 0 | 0
  3 month follow up: 3 days | 0 | 0
  3 month follow up: 2 days | 0 | 0
  3 month follow up: 1 day | 0 | 0
  3 month follow up: 0 days | 0 | 0
  3 month follow up: Unknown or not reported | 1 | 1

3. Primary Outcome: PrEP Adherence Appraisal
Description: One item Medication Adherence question (one item with 5 option scale). "Excellent, Very good, Good, Poor, Very Poor".
Time Frame: one month, three months, three months post intervention
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Intervention | Basic Intervention
Number analyzed (Participants) | 3 | 4
Participants
  1 month: Excellent | 0 | 3
  1 month: Very good | 1 | 0
  1 month: Good | 2 | 0
  1 month: Poor | 0 | 1
  1 month: Very poor | 0 | 0
  1 month: Unknown or not reported | 0 | 0
  3 month: number analyzed (Participants) | 1 | 3
  3 month: Excellent | 0 | 2
  3 month: Very good | 0 | 0
  3 month: Good | 0 | 1
  3 month: Poor | 0 | 0
  3 month: Very poor | 0 | 0
  3 month: Unknown or not reported | 1 | 0
  3 month follow up: number analyzed (Participants) | 1 | 1
  3 month follow up: Excellent | 0 | 0
  3 month follow up: Very good | 0 | 0
  3 month follow up: Good | 0 | 0
  3 month follow up: Poor | 0 | 0
  3 month follow up: Very poor | 1 | 1
  3 month follow up: Unknown or not reported | 0 | 0

4. Secondary Outcome: Coping Self-Efficacy
Description: Assess coping self-efficacy using the Coping Self-Efficacy Scale (13 item scale; 0-10 scale). Zero=cannot do at all,5=moderately certain can do and 10=certain can do. An overall CSE score (from 0 to 130) is created by summing the item ratings, with higher scores indicating higher coping self-efficacy.
Time Frame: Three months, three months post-intervention
Population: Analysis at 3 month and 3 month follow up only includes participants that remained in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Intervention | Basic Intervention
Number analyzed (Participants) | 1 | 3
units on a scale
  3 month | 122 | 101 (28.51)
  3 month follow up: number analyzed (Participants) | 1 | 1
  3 month follow up | 130 | 84

5. Secondary Outcome: Decisional Conflict
Description: Assess decisional conflict with the Ottawa Decisional Conflict Scale. 13 items. 5 responses: Strongly Disagree (1), Disagree (2), Neither Agree or Disagree (3), Agree (4), Strongly Agree (5). Scores are summed and divided by the number of items(13) to produce an overall mean, ranging from 1 to 5. Lower scores indicate lower decisional conflict.
Time Frame: Three months, Three months post intervention
Population: Enhanced group at 3 month (n=1) differs from the overall enhanced group n (17) & basic group at 3 month (n=3) differs from overall basic group n (14) due to implementation barriers that prevented PrEP uptake (e.g., lack of venous access, not returning for doctor appointment), and remaining PrEP adherent (failure to pick up meds, failure to show for appointments). Drop off at 3 month is due to lost to follow up & dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Intervention | Basic Intervention
Number analyzed (Participants) | 1 | 3
units on a scale
  3 month | 5.00 | 4.64 (0.56)
  3 month follow up: number analyzed (Participants) | 1 | 1
  3 month follow up | 5.00 | 4.85

6. Secondary Outcome: PrEP Benefits
Description: 10 items assessed perceived benefits of PrEP. Items are asked on a 0-10 Likert, with 0 = strongly agree, 5 = unsure, 10 = strongly agree. Thus, higher scores indicate greater agreement with that item.
Time Frame: three months, three months post-intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Intervention | Basic Intervention
Number analyzed (Participants) | 1 | 3
units on a scale
  3mo, PrEP can keep me from getting HIV | 9.00 | 9.67 (0.58)
  3mo, Using PrEP would make me feel more in charge of my life | 9.00 | 8.67 (1.53)
  3mo, I would be able to enjoy sex more if I was taking PrEP | 2.00 | 8.67 (1.53)
  3mo, PrEP is easy to take | 10.0 | 10.0 (0)
  3mo, PrEP would not interfere with me injecting or taking drugs | 10.0 | 10.0 (0)
  3mo, I would not have to rely on my partner to use condoms if I was taking PrEP | 10.0 | 4.33 (4.93)
  3mo, I would only have to take one pill a day if I was on PrEP | 10.0 | 10.0 (0)
  3mo, PrEP would let me worry less about HIV | 10.0 | 10.0 (0)
  3mo, I would not have to feel guilty about having fun if I took PrEP | 7.00 | 8.00 (2.00)
  3mo, PrEP is affordable | 10.0 | 9.67 (0.58)
  3mofu, PrEP can keep me from getting HIV: number analyzed (Participants) | 1 | 1
  3mofu, PrEP can keep me from getting HIV | 5.00 | 5.00
  3mofu, Using PrEP would make me feel more in charge of my life: number analyzed (Participants) | 1 | 1
  3mofu, Using PrEP would make me feel more in charge of my life | 5.00 | 5.00
  3mofu, I would be able to enjoy sex more if I was taking PrEP: number analyzed (Participants) | 1 | 1
  3mofu, I would be able to enjoy sex more if I was taking PrEP | 5.00 | 10.00
  3mofu, PreP is easy to take: number analyzed (Participants) | 1 | 1
  3mofu, PreP is easy to take | 5.00 | 10.0
  3mofu, PrEP would not interfere with me injecting or taking drugs: number analyzed (Participants) | 1 | 0
  3mofu, PrEP would not interfere with me injecting or taking drugs | 10.0 |
  3mofu, I would not have to rely on my partner to use condoms if I was taking PrEP: number analyzed (Participants) | 1 | 1
  3mofu, I would not have to rely on my partner to use condoms if I was taking PrEP | 10.0 | 5.0
  3mofu, I would only have to take one pill a day if I Was on PrEP: number analyzed (Participants) | 1 | 1
  3mofu, I would only have to take one pill a day if I Was on PrEP | 10.0 | 10.0
  3mofu, PrEP would let me worry less about HIV: number analyzed (Participants) | 1 | 1
  3mofu, PrEP would let me worry less about HIV | 10.0 | 10.0
  3mofu, I would not have to feel guilty about having fun if I took PrEP: number analyzed (Participants) | 1 | 1
  3mofu, I would not have to feel guilty about having fun if I took PrEP | 10.0 | 7.00
  3mofu, PrEP is affordable: number analyzed (Participants) | 1 | 1
  3mofu, PrEP is affordable | 10.0 | 10.0

7. Secondary Outcome: PrEP Barriers
Description: 12 items assessed perceived barriers to taking PrEP. Items are asked on a 0-10 Likert, with 0 = strongly disagree, 5 = unsure, 10 = strongly agree. Thus, higher score indicates greater agreement with that item.
Time Frame: Three months, Three month post intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Intervention | Basic Intervention
Number analyzed (Participants) | 1 | 3
units on a scale
  3mo, It would be hard for me to take a pill every day | 0.00 | 0.00 (0.00)
  3mo, Taking PrEP would dull my high | 0.00 | 0.00 (0.00)
  3mo, Taking PrEP would cause too many side effects | 0.00 | 2.00 (3.46)
  3mo, I feel healthy so I don't need to take PrEP | 10.0 | 0.00 (0.00)
  3mo, I already protect myself from HIV in other ways (condoms, not sharing needles) | 10.0 | 5.33 (3.51)
  3mo, Even if I take PrEP, I might get HIV anyway | 0.00 | 3.67 (4.04)
  3mo, PrEP only protects against HIV, not other sexually transmitted infections | 10.0 | 10.0 (0.00)
  3mo, My partner might hurt me if they knew I was on PrEP | 0.00 | 0.00 (0.00)
  3mo, I have a lot more worries in my life than getting HIV | 10.0 | 9.00 (1.73)
  3mo, If i started PreP it would be hard to get to the doctor every 3 months | 0.00 | 0.33 (0.58)
  3mo, I don't have a safe place to keep PrEP | 0.00 | 0.00 (0.00)
  3mo, I would be afraid if I had PrEP it would get stolen | 0.00 | 0.00 (0.00)
  3mofu, It would be hard for me to take a pill every day: number analyzed (Participants) | 1 | 1
  3mofu, It would be hard for me to take a pill every day | 5.00 | 0.00
  3mofu, Taking PrEP would dull my high: number analyzed (Participants) | 1 | 1
  3mofu, Taking PrEP would dull my high | 5.00 | 0.00
  3mofu, Taking PrEP would cause too many side effects: number analyzed (Participants) | 1 | 1
  3mofu, Taking PrEP would cause too many side effects | 8.00 | 6.00
  3mofu, I feel healthy so I don't need to take PrEP: number analyzed (Participants) | 1 | 1
  3mofu, I feel healthy so I don't need to take PrEP | 2.00 | 0.00
  3mofu, I already protect myself from HIV in other ways (condoms, not sharing needles): number analyzed (Participants) | 1 | 1
  3mofu, I already protect myself from HIV in other ways (condoms, not sharing needles) | 10.0 | 0.00
  3mofu, Even if I take PrEP, I might get HIV anyway: number analyzed (Participants) | 1 | 1
  3mofu, Even if I take PrEP, I might get HIV anyway | 10.0 | 0.00
  3mofu, PrEP only protects against HIV, not other sexually transmitted infections: number analyzed (Participants) | 1 | 1
  3mofu, PrEP only protects against HIV, not other sexually transmitted infections | 10.0 | 10.0
  3mofu, My partner might hurt me if they knew I was on PrEP: number analyzed (Participants) | 1 | 1
  3mofu, My partner might hurt me if they knew I was on PrEP | 0.00 | 0.00
  3mofu, I have a lot more worries in my life than getting HIV: number analyzed (Participants) | 1 | 1
  3mofu, I have a lot more worries in my life than getting HIV | 5.00 | 5.00
  3mofu, If i started PreP it would be hard to get to the doctor every three months: number analyzed (Participants) | 1 | 1
  3mofu, If i started PreP it would be hard to get to the doctor every three months | 5.00 | 0.00
  3mofu, I don't have a safe place to keep PrEP: number analyzed (Participants) | 1 | 1
  3mofu, I don't have a safe place to keep PrEP | 0.00 | 0.00
  3mofu, I would be afraid if I had PrEP it would get stolen: number analyzed (Participants) | 1 | 1
  3mofu, I would be afraid if I had PrEP it would get stolen | 0.00 | 0.00

8. Secondary Outcome: PrEP Beliefs
Description: 9 items assessed perceived beliefs about PrEP. Items are asked on a 0-10 Likert, with 0 = strongly disagree, 5 = unsure, 10 = strongly agree. Thus, higher score indicates greater agreement with that item.
Time Frame: Three month, Three month post intervention
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Intervention | Basic Intervention
Number analyzed (Participants) | 1 | 3
units on a scale
  3mo, Sex workers need PrEP more than other people | 0.00 | 0.67 (1.16)
  3mo, People who inject drugs need PrEP more than other people | 10.0 | 0.00 (0.00)
  3mo, Gay men need PrEP more than other people | 10.0 | 0.00 (0.00)
  3mo, Trans people need PrEP more than other people | 10.0 | 0.00 (0.00)
  3mo, People from certain races/ethnicities need PrEP more than other people | 0.00 | 0.00 (0.00)
  3mo, PrEP sounds too good to be true | 0.00 | 0.00 (0.00)
  3mo, PrEP makes people think they are invincible (can't get HIV or other sexually transmitted infect | 0.00 | 0.00 (0.00)
  3mo, PrEP is safe and effective for women to use | 10.0 | 9.67 (0.58)
  3mo, I am more likely to take PrEP if I am being paid to take it | 0.00 | 0.00 (0.00)
  3mofu, Sex workers need PrEP more than other people: number analyzed (Participants) | 1 | 1
  3mofu, Sex workers need PrEP more than other people | 10.00 | 0.00
  3mofu, People who inject drugs need PrEP more than other people: number analyzed (Participants) | 1 | 1
  3mofu, People who inject drugs need PrEP more than other people | 10.0 | 0.00
  3mofu, Gay men need PrEP more than other people: number analyzed (Participants) | 1 | 1
  3mofu, Gay men need PrEP more than other people | 10.0 | 0.00
  3mofu, Trans people need PrEP more than other people: number analyzed (Participants) | 1 | 1
  3mofu, Trans people need PrEP more than other people | 10.0 | 0.00
  3mofu, People from certain races/ethnicities need PrEP more than other people: number analyzed (Participants) | 1 | 1
  3mofu, People from certain races/ethnicities need PrEP more than other people | 10.00 | 0.00
  3mofu, PrEP sounds too good to be true: number analyzed (Participants) | 1 | 1
  3mofu, PrEP sounds too good to be true | 0.00 | 0.00
  3mofu, PrEP makes people think they are invincible (can't get HIV or other STIs): number analyzed (Participants) | 1 | 1
  3mofu, PrEP makes people think they are invincible (can't get HIV or other STIs) | 0.00 | 0.00
  3mofu, PrEP is safe and effective for women to use: number analyzed (Participants) | 1 | 1
  3mofu, PrEP is safe and effective for women to use | 10.0 | 10.0
  3mofu, I am more likely to take PrEP if I am being paid to take it: number analyzed (Participants) | 1 | 1
  3mofu, I am more likely to take PrEP if I am being paid to take it | 0.00 | 0.00

ADVERSE EVENTS:
Time Frame: Six months - baseline, intervention (three months), three month followup
Arm/Group | Enhanced Intervention | Basic Intervention
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14

LIMITATIONS AND CAVEATS:
Limitations were: 1.COVID-19 - delayed/disrupted recruitment efforts; 2. 51% of randomized participants were lost-to-follow-up prior to receiving a PrEP prescription due to lack of venous access and lag time getting to see an HIV tester or doctor who were only available certain days due to COVID-19 protocols; 3. Time to engage women for time necessary to complete baseline procedures, HIV testing, and bloodwork as the need to use drugs to avoid withdrawal symptoms superseded study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT03541642/Prot_SAP_ICF_000.pdf